CLINICAL TRIAL: NCT01617122
Title: To Evaluate Bacteriophage OX174 Antigen as a Useful Immunogen in Patients With Immune Deficiency
Brief Title: Evaluate Bacteriophage as a Useful Immunogen in Patients With Primary Immune Deficiency Diseases (PIDD)
Acronym: Bacteriophage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACH 03-0120
Record Dates: First submitted 2010-08-05; First posted 2012-06-12 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Primary Immune Deficiency Diseases
Keywords: PID; PIDD; antibody deficiency; CVID; recurrent infections
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Reinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bacteriophage (Experimental): Subjects receive bacteriophage vaccinations and blood draws
  Interventions: Biological: Bacteriophage OX174

INTERVENTIONS:
Biological: Bacteriophage OX174 — Give first dose of bacteriophage (2 x 109 PFU/kg body weight (0.02 ml/kg)) at visit one. Obtain labs prior to vaccine, 15 minutes, 1 week, 2 weeks, and 4 weeks after vaccine. 6 weeks after 1st vaccine, obtain blood, give 2nd dose of bacteriophage, obtain labs 15 minutes, 1 week, 2 weeks, and 4 weeks after vaccine. Selected patients may receive a tertiary vaccine.

SUMMARY:
This protocol is designed to ascertain whether the bacteriophage 0X174 neoantigen is safe and effective as an antigen used in the evaluation of primary and secondary immune responses. Bacteriophage 0X174 is given intravenously 2 billion PFU/Kg of body weight; small blood specimens of 3-5 ml (about 1 teaspoon) are collected after 15 minutes, 7 days, 14 days, and 28 days. Blood is collected at intervals following the administration of the bacteriophage and the number of phage/ml is determined by the agar overlay method using suspension of E. coli C and serially diluted patient's serum. Phage-specific IgG and IgM are measured by neutralization assay. Capacity of switch from IgM to IgG is determined.

ELIGIBILITY:
Inclusion Criteria:

1. subject/parent or guardian willing to sign consent and adhere to study schedule
2. known or suspected primary immune deficiency

Exclusion Criteria:

1. pregnancy
2. breastfeeding
3. unwilling to sign consent or adhere to study schedule
4. < 2 yrs of age or > 85 yrs of age
5. previous reaction to vaccine

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1995-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of capacity of switch from IgM to IgG. | 12 weeks
  Blood samples are obtained after each immunizition of Bacteriophage.

CONTACTS AND LOCATIONS:
Overall Officials: John W Sleasman, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, St. Petersburg, Florida, United States